CLINICAL TRIAL: NCT05257291
Title: Melatonin and Essential Arterial Hypertension
Brief Title: Study MIPAE - Melatonin and Essential Arterial Hypertension
Acronym: MIPAE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Rita Rezzani, PhD, Full Professor of Human Anatomy, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 2717
Record Dates: First submitted 2021-10-06; First posted 2022-02-25 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Melatonin; Antioxidant; Antihypertensive; Cardiovascular System
MeSH Terms: conditions — Essential Hypertension | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Group of essential hypertensive patients who have received no additional therapies in addition to their established treatment plan (each patient was on specific antihypertensive therapy that has not been changed).
- Melatonin treated group (Active Comparator): Group of essential hypertensive patients who have received additional therapies consisting in 1 mg/day of melatonin for 1 year, in addition to their established treatment plan.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Supplementation with 1 mg/day of melatonin for 1 year
  Arms: Melatonin treated group

SUMMARY:
Study MIPAE - Melatonin and essential arterial hypertension.

Study with dietary supplement, prospective and monocentric (randomized control trial). 1 mg/day of melatonin has been administered for one year to a group of patients suffering from essential hypertension (from at least one year) and who are already on antihypertensive therapy. This group has been compared with as many hypertensive patients on antihypertensive therapy to whom melatonin has not been administered. Each of the participants have been evaluated at the beginning of the study and after one year considering:

* systolic and diastolic blood pressure;
* echocardiographic values (Vivid Q, GE Healthcare);
* applanation tonometry (SphygmoCor, AtCor Medical);
* peripheral arterial tonometry (EndoPAT-2000, Itamar);
* melatonin levels and total circulating antioxidant capacity after peripheral venous blood sampling.

The aim of the study was to evaluate the antioxidant and vasoprotective effects of melatonin, evaluating both plasma changes and directly studying the possibility of a real remodeling and improvement of cardiac structures.

DETAILED DESCRIPTION:
Hypertension is a pathological condition characterized by a constant and not occasional increase in systolic and diastolic blood pressure values. This pathology represents one of the most important public health problems in industrialized countries, as it affects more than 25-30% of the adult population and can cause serious and even fatal complications. It is in fact considered the major risk factor of mortality and pathological effect at cardiovascular, encephalic and renal level.

The classification of hypertension suggested by the ESC/ESH Guidelines defines diastolic blood pressure (PAD) values of 80-84 mmHg and systolic blood pressure (PAS) values of 120-129 mmHg as "normal" in a healthy adult. Blood pressure values between 90-99 mmHg (PAD) and 140-159 mmHg (PAS) define grade 1 hypertension.Between 100-109 mmHg (PAD) and 160-179 mmHg (PAS) define grade 2 hypertension. For values above 110 mmHg (PAD) and 180 mmHg (PAS), determine grade 3 hypertension (after 60 years of age slightly higher values are accepted). Although many antihypertensive drug therapies exist today, patients often show a lack of response to pharmacological treatment due to numerous factors of both genetic and environmental nature that contribute to determine the clinical picture and the poor response to the set therapeutic regime. Recent studies aimed at clarifying the pathophysiology of resistant hypertension are highlighting new pathophysiological mechanisms potentially involved in the genesis of this clinical condition. Since essential hypertension and vascular and cardiac dysfunctions seem to be closely related, the identification of molecules/substances that can at least help to reduce the alterations induced by the pathogenetic process of essential hypertension is a priority. In recent years, melatonin has shown important and interesting antihypertensive therapeutic potential. It has also been demonstrated by some authors of this project, in an animal model of arterial hypertension, that melatonin, thanks to its antioxidant properties, is able to regress structural alterations of both the aorta and small mesenteric resistance arteries in an animal model of arterial hypertension.

It is therefore necessary to investigate, also in humans, the correlation among essential arterial hypertension, levels of circulating melatonin and onset of cardiovascular events.

Furthermore, it is of fundamental importance to remember that, to date, following treatment with melatonin, even at high doses, show only rare and minimal adverse effects, including daytime drowsiness, dizziness and headaches.

The aim of the study was, therefore, to evaluate the antihypertensive, antioxidant and vasoprotective effects of melatonin in adult patients suffering from at least 1 year essential hypertension and in antihypertensive therapy. In a broad sense, the aim will be to contribute to current knowledge in terms of effective treatment and reduced impact of cardiovascular changes related to hypertension.

To do this, a total of 23 adult patients (mean age 54 years old) suffering from essential arterial hypertension and undergoing concurrent antihypertensive therapy were enrolled by the Cardiology Unit of the Spedali Civili di Brescia (Italy). The participants were randomly divided into a group to which melatonin was administered orally (1 mg/day for one year - "melatonin" group). This group of patients was then compared with a group of hypertensive patients on antihypertensive therapy who did not take melatonin ("control" group). In particular, patients with essential hypertension for at least 1 year were selected and enrolled.

With regard to the number of samples, reference has been made to recent studies conducted at our Institute. The sample size (alpha 0.05, power 80%) needed to catch a 2 tissue strain modification of the ascending aorta is 6.2% of the longitudinal 2D strain of the left ventricle 21, 0.1 of VAC is 10, 0.25 of RH-PAT index 17, 0.5 m/s in cfPWV is 12. In addition, patients after enrolment have been randomized 1:1 in the two groups; randomization by random number generation minimizes selection prejudices/errors in subdivising into groups and allows to better evaluate the possible effects of melatonin treatment on hypertensive patients (on antihypertensive therapy) compared to hypertensive patients (on antihypertensive) therapy who have not taken melatonin, while the other variables and the analysis to be performed have been kept constant.

All patients with essential hypertension (in antihypertensive therapy) enrolled in the study received the informed consent document and the information document together with clear and understandable explanations/information about the study. In addition, the investigating physician is available to enlisted patients for all necessary information and also for any subsequent questions/curiosities, as well as for the reporting of any adverse effects that he or she undertakes to notify promptly.

In addition, the supply of melatonin tablets required for 30 ± 3 days of treatment (35 tablets of 1 mg melatonin) have been delivered by the investigating physician only to patients enrolled in the "melatonin" group at the time of enrolment and for the following 11 months of the trial.

At the time of enrolment, the investigator has also provided all enlisted subjects a diary on which to record the time of melatonin intake (only for the "melatonin" group), the number of hours of sleep at night, the systolic and diastolic blood pressure values measured weekly by the patient himself and the onset of any adverse effects. At the end of the study, the investigator collected the diaries of all patients enrolled in the study in order to analyze and archive the data together with the evaluation of the previous medical history.

At the beginning of the study and after one year, the patients were evaluated during a medical examination considering:

* blood pressure (weekly evaluation carried out by the patient and monthly check-up carried out by the investigating doctor during meetings with the patient);
* heart rate;
* endothelial parameters: RHI, LnRHI, peripheral AIx@75;
* arterial stiffness parameters: central blood pressure, AIx@75 radial, cfPWV, SEVR;
* echocardiographic parameters: dimensions of atria and ventricles, stenosis and valve insufficiencies, systolic function VS (FE) and VD (TAPSE, FAC, S' TSI), diastolic function VS and VD (E/A, DT, E/E', E'/A'), dimensions and elastic properties of the ascending aorta (compliance, distensibility, stiffness index, elastic modulus of Peterson, PWV, M-mode strain, tissue strain), elongated aortic (Ea) and ventricular telediastolic sinintra (Ees), ventricular-arterial coupling (VAC=Ea/Ees), 2D longitudinal/radial/circonferential strain of VS, longitudinal strain of VD and left atrium (LAA and LAS), torsion of VS;
* laboratory parameters: blood melatonin levels and total circulating antioxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian race;
* Age 40-50;
* Signed written informed consent
* Normal weight;
* Blood pressure: PAD >90 mmHg and PAS >140 mmHg;
* Blood pressure in the above mentioned range from at least 1 years
* Fasting blood sugar < 100 mg/dL;
* Total cholesterol < 200 mg/dL and triglycerides < 150 mg/dL;
* Intake of antihypertensive therapies (except nitrates, statins and β-blockers);
* Non-smoking;
* No night shift workers (at least in the last 3 months before recruitment);
* With a regular sleep/wake rhythm;
* No pregnant/nursing women.

Exclusion Criteria:

* Blood pressure: PAD <90 mmHg and PAS <140 mmHg
* Heart disease of any kind;
* Autoimmune or rheumatological or vascular diseases other than essential hypertension;
* Anti-hypertensive therapies with nitrates, statins or β-blockers;
* Pregnancy/nursing;
* < 40 or > 50 years;
* Worker with night shifts (for a period of less than 3 months before recruitment);
* Continuous irregular sleep/wake rhythm.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure. | Baseline.
  Value of ambulatory blood pressure obtained from the mean of three different misurations.
Heart rate. | Baseline.
  Ambulatory recorder of the heart rate of the patient.
Endothelial parameters. | Baseline.
  PAT signals were obtained using the EndoPAT-2000 device, which has been vali-dated and used previously to assess peripheral arterial tone in other populations. Endothelial function is measured via a reactive hyper-emia (RH) protocol: it consists of a 5 minutes baseline mea-surement, after which a blood pressure cuff on the test arm isinflated to 60 mm Hg above baseline systolic BP or at least200 mm Hg for 5 minutes. After 5 minutes, the cuff is deflated, and the PAT tracing isrecorded for a further 5 minutes. The cal-culated ratio is called RH-PAT index or RH index (RHI).
Arterial stiffness parameters. | Baseline.
  The radial artery waveform was recorded using the SphygmoCor system. The tip of the tonometer was pressed gently against the radial artery at the site of maximum pulsation at the wrist. This micromanometer precisely records pressure within the artery. he augmentation pressure is defined as the height of the late systolic peak above the inflection point. Augmentation index is expressed as a percentage of PPAO. Augmentation index is a measure of the stiffness of the arterial walls, namely pulsatile load. Because there is a linear relationship between it and heart rate (HR), augmentation index was standardized to a HR of 75 bpm (AIx@75).
Echocardiographic parameters. | Baseline.
  Bi-dimensional transthoracic echocardiographic examinations were performed using Vivid 9 and Vivid Q (GE Medical HealthCare, USA) with a probe of 3.5 MHz, to assess LV dimensions and systolic function, according to the guidelines. The main points were: the dimensions of atria and ventricles, stenosis and valve insufficiencies, systolic and diastolic function VS and VD, Dimensions and elastic properties of the ascending aorta (compliance, distensibility, stiffness index, elastic modulus of Peterson, PWV, M-mode strain, tissue strain).
Plasmatic melatonin levels. | Baseline.
  Obtained with ELISA laboratory test.
Total circulating antioxidant capacity in plasma. | Baseline.
  Obtained with ELISA laboratory test.
Blood pressure. | 1 year.
  Ambulatory blood pressure obtained from the mean of three different misurations.
Heart rate. | 1 year.
  Ambulatory recorder of the heart rate of the patient.
Endothelial parameters. | 1 year.
  PAT signals were obtained using the EndoPAT-2000 device, which has been vali-dated and used previously to assess peripheral arterial tone in other populations. Endothelial function is measured via a reactive hyper-emia (RH) protocol: it consists of a 5 minutes baseline mea-surement, after which a blood pressure cuff on the test arm isinflated to 60 mm Hg above baseline systolic BP or at least200 mm Hg for 5 minutes. After 5 minutes, the cuff is deflated, and the PAT tracing isrecorded for a further 5 minutes. The cal-culated ratio is called RH-PAT index or RH index (RHI).
Arterial stiffness parameters. | 1 year.
  The radial artery waveform was recorded using the SphygmoCor system. The tip of the tonometer was pressed gently against the radial artery at the site of maximum pulsation at the wrist. This micromanometer precisely records pressure within the artery. he augmentation pressure is defined as the height of the late systolic peak above the inflection point. Augmentation index is expressed as a percentage of PPAO. Augmentation index is a measure of the stiffness of the arterial walls, namely pulsatile load. Because there is a linear relationship between it and heart rate (HR), augmentation index was standardized to a HR of 75 bpm (AIx@75).
Echocardiographic parameters. | 1 year.
  Bi-dimensional transthoracic echocardiographic examinations were performed using Vivid 9 and Vivid Q (GE Medical HealthCare, USA) with a probe of 3.5 MHz, to assess LV dimensions and systolic function, according to the guidelines. The main points were: the dimensions of atria and ventricles, stenosis and valve insufficiencies, systolic and diastolic function VS and VD, Dimensions and elastic properties of the ascending aorta (compliance, distensibility, stiffness index, elastic modulus of Peterson, PWV, M-mode strain, tissue strain).
Plasmatic melatonin levels. | 1 year.
  Obtained with ELISA laboratory test.
Total circulating antioxidant capacity in plasma. | 1 year.
  Obtained with ELISA laboratory test.

CONTACTS AND LOCATIONS:
Locations (1):
- Anatomy and Physiopathology Division, Department of Experimental and Clinical Sciences, University of Brescia (Italy), Viale Europa 11, 25123 Brescia, Italy, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Scientific publication in an international peer-reviewed journal
Time Frame: illimited
Access Criteria: upon request

REFERENCES:
- [Background] Acuna-Castroviejo D, Escames G, Venegas C, Diaz-Casado ME, Lima-Cabello E, Lopez LC, Rosales-Corral S, Tan DX, Reiter RJ. Extrapineal melatonin: sources, regulation, and potential functions. Cell Mol Life Sci. 2014 Aug;71(16):2997-3025. doi: 10.1007/s00018-014-1579-2. Epub 2014 Feb 20. PMID 24554058
- [Background] Agabiti-Rosei C, De Ciuceis C, Rossini C, Porteri E, Rodella LF, Withers SB, Heagerty AM, Favero G, Agabiti-Rosei E, Rizzoni D, Rezzani R. Anticontractile activity of perivascular fat in obese mice and the effect of long-term treatment with melatonin. J Hypertens. 2014 Jun;32(6):1264-74. doi: 10.1097/HJH.0000000000000178. PMID 24751595
- [Background] Andersen LP, Gogenur I, Rosenberg J, Reiter RJ. The Safety of Melatonin in Humans. Clin Drug Investig. 2016 Mar;36(3):169-75. doi: 10.1007/s40261-015-0368-5. PMID 26692007
- [Background] Arangino S, Cagnacci A, Angiolucci M, Vacca AM, Longu G, Volpe A, Melis GB. Effects of melatonin on vascular reactivity, catecholamine levels, and blood pressure in healthy men. Am J Cardiol. 1999 May 1;83(9):1417-9. doi: 10.1016/s0002-9149(99)00112-5. PMID 10235107
- [Background] Bonetti PO, Lerman LO, Lerman A. Endothelial dysfunction: a marker of atherosclerotic risk. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):168-75. doi: 10.1161/01.atv.0000051384.43104.fc. PMID 12588755
- [Background] Cagnacci A, Arangino S, Angiolucci M, Maschio E, Longu G, Melis GB. Potentially beneficial cardiovascular effects of melatonin administration in women. J Pineal Res. 1997 Jan;22(1):16-9. doi: 10.1111/j.1600-079x.1997.tb00297.x. PMID 9062865
- [Background] Cagnacci A, Arangino S, Angiolucci M, Melis GB, Facchinetti F, Malmusi S, Volpe A. Effect of exogenous melatonin on vascular reactivity and nitric oxide in postmenopausal women: role of hormone replacement therapy. Clin Endocrinol (Oxf). 2001 Feb;54(2):261-6. doi: 10.1046/j.1365-2265.2001.01204.x. PMID 11207642
- [Background] Chen CH, Fetics B, Nevo E, Rochitte CE, Chiou KR, Ding PA, Kawaguchi M, Kass DA. Noninvasive single-beat determination of left ventricular end-systolic elastance in humans. J Am Coll Cardiol. 2001 Dec;38(7):2028-34. doi: 10.1016/s0735-1097(01)01651-5. PMID 11738311
- [Background] Conti A, Conconi S, Hertens E, Skwarlo-Sonta K, Markowska M, Maestroni JM. Evidence for melatonin synthesis in mouse and human bone marrow cells. J Pineal Res. 2000 May;28(4):193-202. doi: 10.1034/j.1600-079x.2000.280401.x. PMID 10831154
- [Background] Favero G, Rodella LF, Reiter RJ, Rezzani R. Melatonin and its atheroprotective effects: a review. Mol Cell Endocrinol. 2014 Feb 15;382(2):926-37. doi: 10.1016/j.mce.2013.11.016. Epub 2013 Nov 28. PMID 24291636
- [Background] Goor DA, Sheffy J, Schnall RP, Arditti A, Caspi A, Bragdon EE, Sheps DS. Peripheral arterial tonometry: a diagnostic method for detection of myocardial ischemia induced during mental stress tests: a pilot study. Clin Cardiol. 2004 Mar;27(3):137-41. doi: 10.1002/clc.4960270307. PMID 15049379
- [Background] Hardeland R, Cardinali DP, Srinivasan V, Spence DW, Brown GM, Pandi-Perumal SR. Melatonin--a pleiotropic, orchestrating regulator molecule. Prog Neurobiol. 2011 Mar;93(3):350-84. doi: 10.1016/j.pneurobio.2010.12.004. Epub 2010 Dec 28. PMID 21193011
- [Background] Intengan HD, Schiffrin EL. Vascular remodeling in hypertension: roles of apoptosis, inflammation, and fibrosis. Hypertension. 2001 Sep;38(3 Pt 2):581-7. doi: 10.1161/hy09t1.096249. PMID 11566935
- [Background] Kawasaki T, Sasayama S, Yagi S, Asakawa T, Hirai T. Non-invasive assessment of the age related changes in stiffness of major branches of the human arteries. Cardiovasc Res. 1987 Sep;21(9):678-87. doi: 10.1093/cvr/21.9.678. PMID 3328650
- [Background] Laurent S, Boutouyrie P. The structural factor of hypertension: large and small artery alterations. Circ Res. 2015 Mar 13;116(6):1007-21. doi: 10.1161/CIRCRESAHA.116.303596. PMID 25767286
- [Background] Lundberg MS, Crow MT. Age-related changes in the signaling and function of vascular smooth muscle cells. Exp Gerontol. 1999 Jul;34(4):549-57. doi: 10.1016/s0531-5565(99)00036-4. PMID 10817810
- [Background] Meissner A, Minnerup J, Soria G, Planas AM. Structural and functional brain alterations in a murine model of Angiotensin II-induced hypertension. J Neurochem. 2017 Feb;140(3):509-521. doi: 10.1111/jnc.13905. Epub 2016 Dec 21. PMID 27874975
- [Background] Nawaz W, Khan FU, Khan MZ, Gang W, Yang M, Liao X, Zhang L, Ihsan AU, Khan A, Han L, Zhou X. Exo-organoplasty interventions: A brief review of past, present and future directions for advance heart failure management. Biomed Pharmacother. 2017 Apr;88:162-172. doi: 10.1016/j.biopha.2017.01.048. Epub 2017 Jan 16. PMID 28103510
- [Background] Oktay AA, Lavie CJ, Milani RV, Ventura HO, Gilliland YE, Shah S, Cash ME. Current Perspectives on Left Ventricular Geometry in Systemic Hypertension. Prog Cardiovasc Dis. 2016 Nov-Dec;59(3):235-246. doi: 10.1016/j.pcad.2016.09.001. Epub 2016 Sep 8. PMID 27614172
- [Background] Orabona R, Sciatti E, Vizzardi E, Bonadei I, Valcamonico A, Metra M, Frusca T. Endothelial dysfunction and vascular stiffness in women with previous pregnancy complicated by early or late pre-eclampsia. Ultrasound Obstet Gynecol. 2017 Jan;49(1):116-123. doi: 10.1002/uog.15893. PMID 26918484
- [Background] Rezzani R, Porteri E, De Ciuceis C, Bonomini F, Rodella LF, Paiardi S, Boari GE, Platto C, Pilu A, Avanzi D, Rizzoni D, Agabiti Rosei E. Effects of melatonin and Pycnogenol on small artery structure and function in spontaneously hypertensive rats. Hypertension. 2010 Jun;55(6):1373-80. doi: 10.1161/HYPERTENSIONAHA.109.148254. Epub 2010 Apr 26. PMID 20421515
- [Background] Rizzoni D, Porteri E, De Ciuceis C, Boari GE, Zani F, Miclini M, Paiardi S, Tiberio GA, Giulini SM, Muiesan ML, Castellano M, Rosei EA. Lack of prognostic role of endothelial dysfunction in subcutaneous small resistance arteries of hypertensive patients. J Hypertens. 2006 May;24(5):867-73. doi: 10.1097/01.hjh.0000222756.76982.53. PMID 16612248
- [Background] Sarkar T, Singh NP. Epidemiology and Genetics of Hypertension. J Assoc Physicians India. 2015 Sep;63(9):61-98. PMID 27608868
- [Background] Scuteri A, Nilsson PM, Tzourio C, Redon J, Laurent S. Microvascular brain damage with aging and hypertension: pathophysiological consideration and clinical implications. J Hypertens. 2011 Aug;29(8):1469-77. doi: 10.1097/HJH.0b013e328347cc17. PMID 21577138
- [Background] Sorriento D, Santulli G, Del Giudice C, Anastasio A, Trimarco B, Iaccarino G. Endothelial cells are able to synthesize and release catecholamines both in vitro and in vivo. Hypertension. 2012 Jul;60(1):129-36. doi: 10.1161/HYPERTENSIONAHA.111.189605. Epub 2012 Jun 4. PMID 22665130